CLINICAL TRIAL: NCT05325905
Title: Analysis of Gingival Crevicular Fluid IL-1β, IL-10, IL-36γ Cytokine Levels in Gingivitis and Periodontitis Patients
Brief Title: Analysis of Gingival Crevicular Fluid
Acronym: GCF
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehtikar Gursel, Prof.Dr, Bezmialem Vakif University
Other Study IDs: 2014/01
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Periodontal Diseases
Keywords: pathogenesis; Gingival crevicular fluid; cytokine
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: bleeding on probing (BoP) ≤ 10% of the sites, probing depth (PD) ≤ 3 mm and no indication of clinical attachment level (CAL) or radiographic bone loss
  Interventions: Diagnostic Test: Gingival crevicular fluid sampling
- Gingivitis: gingival inflammation (BoP ≥ 10% of the sites, red-blue discoloration of the gingiva and edema) PD ≤ 4 mm and no clinical attachment or radiographic bone loss
  Interventions: Diagnostic Test: Gingival crevicular fluid sampling
- Periodontitis: PD ≤ 5 mm, radiographic bone loss, and 3-4 mm CAL in at least 30% of the sites
  Interventions: Diagnostic Test: Gingival crevicular fluid sampling

INTERVENTIONS:
Diagnostic Test: Gingival crevicular fluid sampling — GCF sampling and clinical periodontal measurements were performed

SUMMARY:
The purpose of this study was to investigate and compare GCF interleukin-1β (IL-1β), interleukin-10 (IL-10), interleukin-36γ (IL-36γ) levels in patients with healthy (H), gingivitis (G) and chronic periodontitis (CP) status.

DETAILED DESCRIPTION:
Gingival crevicular fluid (GCF) is formed when fluid exudes from the vessels of the microcirculation into the inflamed periodontal tissue and into the sulcus or pocket. As the fluid traverses the inflamed tissue, it is thought to pick up enzymes and other molecules that participate in the destructive process, as well as products of cell and tissue degradation. Efforts to develop diagnostic tests based on host factors have been focused almost entirely on analysis of GCF.

The purpose of this study was to investigate and compare GCF interleukin-1β (IL-1β), interleukin-10 (IL-10), interleukin-36γ (IL-36γ) levels in patients with healthy (H), gingivitis (G) and chronic periodontitis (CP) status.

Systemically healthy and non-smokers 80 participants (30 males and 50 females) who were selected from among admitting to Dentistry Faculty of Selcuk University were included in this study. Clinical periodontal parameters were recorded and GCF samples were obtained. Samples were stored in -80 ˚C until analysis with Enzyme-Linked ImmunoSorbent Assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* non-smokers,
* presence of at least 20 teeth in the mouth

Exclusion Criteria:

* receiving periodontal therapy in the last 6 months;
* receiving antibiotics or anti-inflammatory drugs in the last 6 months;
* currently pregnant or breastfeeding
* using a removable partial denture and removable or fixed orthodontic appliances.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were selected from among admitting to Dentistry Faculty of Selcuk University.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Interleukin-36γ (IL-36γ) levels in GCF | Baseline
  GCF samples were obtained from one interproximal site in each quadrant

SECONDARY OUTCOMES:
Probing depth (PD) | Baseline
  PD; from six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual locations) of each tooth other than third molars.
Clinical attachment level (CAL) | Baseline
  CAL; from six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual locations) of each tooth other than third molars.
Bleeding on Probing (BoP) | Baseline
  BoP, from six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual locations) of each tooth other than third molars
IL-10 and IL-1β levels in GCF | Baseline
  GCF samples were obtained from one interproximal site in each quadrant
Plaque Index (PI) | Baseline
  PI; from six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual locations) of each tooth other than third molars
Gingival Index (GI) | Baseline
  GI; from six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual locations) of each tooth other than third molars

CONTACTS AND LOCATIONS:
Overall Officials: Mehtikar Gürsel, Principal Investigator — Bezmialem University

IPD SHARING:
Plan to Share IPD: No
Results will be shared if requested